CLINICAL TRIAL: NCT02017561
Title: Metformin in the Diastolic Dysfunction of Metabolic Syndrome: MET-DIME Trial
Brief Title: Metformin in the Diastolic Dysfunction of Metabolic Syndrome
Acronym: MET-DIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Ricardo Ladeiras-Lopes, Dr. Ricardo Ladeiras-Lopes, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01.00240
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome X; Diastolic Dysfunction; Insulin Resistance
Keywords: Diastolic dysfunction; Metabolic syndrome; Metformin
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Counseling (Active Comparator): Written and individualized information during the interview in all clinic visits, emphasizing the importance of regular moderate-intensity physical activity and healthy diet.
  Interventions: Behavioral: Lifestyle Counseling
- Metformin + Lifestyle Counseling (Experimental): Metformin: maximum dose of 1000mg twice daily. Lifestyle counseling: Written and individualized information during the interview in all clinic visits, emphasizing the importance of regular moderate-intensity physical activity and healthy diet.
  Interventions: Behavioral: Lifestyle Counseling; Drug: Metformin

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Written and individualized information during the interview in all clinic visits, emphasizing the importance of a healthy lifestyle, engaging on regular moderate-intensity physical activity and eating an healthy diet.
Drug: Metformin — Metformin treatment titrated to a maximum dose of 1000mg twice a day. Metformin treatment will start with 500mg at breakfast during the first week and, if well tolerated, increased to 500mg twice a day (breakfast and dinner) in the second week, 1000mg at breakfast and 500mg at dinner in the third week and finally for the target dose of 1000mg twice a day.
  Other Names: Risidon; Glucophage
  Arms: Metformin + Lifestyle Counseling

SUMMARY:
Metabolic syndrome (MS) is a cluster of risk factors for cardiovascular disease with increasing prevalence worldwide and insulin resistance is central to its pathophysiology and multi-organ deleterious effects. One of the most affected organs, the heart, undergoes a remodeling process with an increase in fibrous tissue that impairs global cardiac function. Considering that myocardial fibrosis increases myocardial stiffness, one important determinant of diastolic function, it probably contributes decisively to subclinical left ventricular diastolic dysfunction (DD) and heart failure with preserved ejection fraction in patients with MS.

Since insulin resistance is a dominant player in the pathophysiology of MS, improvement of the metabolic profile of these patients with metformin might be associated with favorable remodeling of myocardial structure and an improvement in myocardial function. Metformin is a widely used drug to treat type 2 diabetes mellitus and is considered an option in the treatment of high-risk non-diabetic patients with MS, in addition to lifestyle counseling including a healthy diet and physical activity.

In this way, we aim to: i) assess if treating non-diabetic patients with MS and DD with metformin in addition to lifestyle counseling decreases cardiac fibrosis and improves diastolic function and assess its impact in functional capacity and health-related quality of life (HRQoL); ii) evaluate if biomarkers of cardiac remodeling and inflammation are predictive factors of response to metformin treatment in these patients.

This is a prospective, randomized, open-label, blinded-endpoint (PROBE) trial (scheduled follow-up of 24 months) with 2 arms: lifestyle counseling only and lifestyle counseling plus metformin (maximum dose of 1000mg twice daily).

The primary endpoint will be change in change in mean of septal and lateral early diastolic mitral annular velocities (E') (at the end of the 24 months of follow-up).

The secondary endpoints will include a composite of major cardiovascular events; diastolic function parameters at rest; plasma levels of insulin, glucose, insulin resistance index, NTproBNP, high-sensitivity C-reactive protein, tumor necrosis factor-α (TNFα), tissue inhibitor of matrix metalloproteinase type 1 (TIMP1) and growth differentiation factor-15 (GDF-15); functional capacity; epicardial, pericardial and abdominal adipose tissue volumes, and coronary calcium score; HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic adults aged between 40 and 64 years fulfilling the American Heart Association/National Heart, Lung and Blood Institute diagnostic criteria of metabolic syndrome (at least 3 of the following: waist circumference ≥102 cm (males) or ≥88 cm (females); fasting triglycerides≥150 mg/dL or on drug therapy for decreasing triglycerides; fasting HDL-cholesterol ˂40 mg/dL (males) or ˂50 mg/dL (females) or on drug therapy for increase HDL-c; systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg or on antihypertensive drug therapy; fasting glycemia≥100 mg/dL
* Echocardiographic evidence of left ventricle diastolic dysfunction at rest (mean E'˂10,2 cm/s if 40-59 years and ˂7,2 cm/s if 60-64 years).

Exclusion Criteria:

* diagnosis of diabetes mellitus according to the American Diabetes Association criteria;
* previous diagnosis of ischemic heart disease;
* moderate or severe cardiac valvular disease;
* left ventricle ejection fraction lower than 50%
* pericardial disease;
* uncontrolled atrial or ventricular tachyarrhythmias;
* chronic kidney disease (estimated creatinine clearance lower than 60 mL/min);
* significant liver disease (aspartate aminotransferase or alanine aminotransferase equal or above 2.5 times the upper limit of normal);
* females who are pregnant, planning to become pregnant or who admit sexual activity without appropriate contraception;
* lactation;
* unable to perform cardiopulmonary exercise test;
* recent (less than 1 month) change in drug therapy.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in mean early diastolic mitral annular velocity (cm/s) | Baseline, 6,12 and 24 months
  Change in mean of septal and lateral early diastolic mitral annular velocities (E'), assessed by tissue doppler echocardiography

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 and 24 months
  Composite outcome of major cardiovascular events: nonfatal myocardial infarction, nonfatal stroke, death judged to be due to cardiovascular causes, hospitalization for heart failure, angina confirmed by ischemic changes on exercise tolerance testing or by clinically significant obstruction on coronary angiography or need for revascularization with angioplasty or coronary-artery bypass grafting.
Diastolic echocardiographic parameters | Baseline, 6, 12, 24 months
  E/E´ ratio, isovolumetric relaxation time (IVRT), E/A ratio, mitral deceleration time, grade of diastolic dysfunction according to the consensus document of the American Society of Echocardiography and European Society of Echocardiography, strain rate during isovolumetric relaxation (SR-IVR) and E/SR-IVR ratio.
Plasma levels of inflammatory and metabolic biomarkers | Baseline, 6, 12, 24 months
  Plasma levels of insulin, glucose, insulin resistance index, NTproBNP, high-sensitivity C-reactive protein, TNFα, TIMP1 e GDF-15 (growth differentiation factor 15).
Functional capacity during cardiopulmonary exercise test | Baseline, 12, 24 months
  Functional capacity during cardiopulmonary exercise test: all patients will perform a symptom-limited treadmill exercise testing according to modified Bruce protocol, with simultaneous respiratory gas analysis. Peak oxygen uptake, anaerobic threshold and ventilatory efficiency will be determined.
Epicardial, pericardial and abdominal adipose tissue volumes | Baseline, 24 months
  Cardiac multidetector CT without contrast administration to measure epicardial, pericardial and abdominal adipose tissue volumes
Coronary artery calcium quantification | Baseline, 24 months
  Cardiac multidetector CT without contrast administration to assess coronary artery calcification (calcium score)
Healthcare related quality of life | Baseline, 12, 24 months
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) will be used to assess general health status and HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ladeiras-Lopes, MD, Principal Investigator — Department of Physiology and Cardiothoracic Surgery, Faculty of Medicine of the University of Porto; Adelino F Leite-Moreira, MD,PhD,FETCS, Study Chair — Department of Physiology and Cardiothoracic Surgery, Faculty of Medicine of the University of Porto; Vasco Gama, MD, Study Chair — Department of Cardiology, Gaia/Espinho Hospital Centre
Locations (1):
- Gaia/Espinho Hospital Centre, Vila Nova de Gaia, Portugal